CLINICAL TRIAL: NCT00621309
Title: Phase I Clinical Trial to Evaluate the Efficacy of Sulforaphane as an Antagonist to Human PXR-mediated Drug-drug Interactions
Brief Title: Sulforaphane as an Antagonist to Human PXR-mediated Drug-drug Interactions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Fred Hutchinson Cancer Center (Other); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, David Eaton, Professor, Environmental and Occupational Health Sciences, University of Washington
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 33109; NIH grant: 1R01GM079280-01A1;; 07-9114-A01
Record Dates: First submitted 2008-02-12; First posted 2008-02-22 (Estimated); Results first posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-08

CONDITIONS: Adverse Drug Interactions
Keywords: drug interactions; cytochrome P4503A4; Pregnane X-receptor; induction; drug metabolism
MeSH Terms: interventions — Rifampin; rifamycin SV; sulforaphane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): Subjects are given 300 mg / 7 days of rifampicin to induce CYP3A4. Midazolam clearance is measured on the 8th day.
  Interventions: Drug: Rifampicin
- 2 (Active Comparator): Sulforaphane (SFN), a natural product derived from broccoli sprouts, is utilized as a putative inhibitor of ligand (Rifampin) activation of the Pregnane X-receptor. In this arm, both SFN (putative inhibitor of ligand binding to PXR) and Rifampin (strong activating ligand of PXR) are given together.
  Interventions: Dietary Supplement: sulforaphane plus rifampicin
- 3 (Active Comparator): This arm involves the administration of Sulforaphane (SFN) alone, in the absence of the PXR ligand, rifampicin. The hypothesis is that SFN will have no effect on the expression of PXR-regulated genes. Alternatively, it is possible that SFN could inhibit as yet unidentified endogenous ligands to the PXR receptor, thereby causing down-regulations of genes regulated wholely or in part by PXR. SFN is administered as a broccoli sprout extract at a dose rate of 75 mg (~420 umoles) per day for 7 days.
  Interventions: Dietary Supplement: sulforaphane alone

INTERVENTIONS:
Drug: Rifampicin — Rifampicin, an antibiotic used to treat TB, is administered at a dose of 300 mg day x 7 days to induce CYP3A5.
  Other Names: Rifampin; rifamycin; Rimactane; Rifadin
  Arms: 1
Dietary Supplement: sulforaphane plus rifampicin — Sulforaphane (SFN) is an isothiocyanate derived from the plant phytochemical, glucoraphinin. It appears to inhibit ligand binding to the ligand activated nuclear transcription factor, Pregnane X-Receptor (PXR). This arm tests the hypothesis that SFN can block ligand binding to the PXR, thereby inhibiting transcriptional activation of PXR-regulated genes. Sulforaphane is administered daily for 7 days as a broccoli sprout extract, at a dose rate of 75 mg (~420 umoles)per day for 7 days. Rifampicin is also administered once per day at a dose rate of 300 mg/day for 7 days.
  Other Names: sulforaphane: glucoraphinin (precursor); 1-Isothiocyanato-4-methylsulfinyl-butane; Rifampicin: Rifampin, Rifadin, Rimactane
  Arms: 2
Dietary Supplement: sulforaphane alone — Sulforaphane (SFN) is an isothiocyanate derived from the plant phytochemical, glucoraraphinin. It appears to inhibit ligand binding to the ligand activated nuclear transcription factor, Pregnane X-Receptor (PXR). This arm tests the hypothesis that SFN can block ligand binding to the PXR, thereby inhibiting transcriptional activation of PXR-regulated genes
  Other Names: 1-isothiocyanato-4-(methylsulphinyl)butane
  Arms: 3

SUMMARY:
Adverse drug-drug interactions (DDIs) are responsible for approximately 3% of all hospitalizations in the US, perhaps costing more than $1.3 billion per year. One of the most common causes of DDIs is the when one drug alters the metabolism of another. A key enzyme in the liver and intestine, called "cytochrome P450 3A4 (CYP3A4) is generally considered to be the most important drug metabolizing enzyme. The gene for CYP3A4 can be 'turned on' by the presence of certain other drugs, resulting in much higher levels of CYP3A4 in the liver and intestine. Thus, when a drug that induces CYP3A4 is given with or before another drug that is metabolized by 3A4, a 'drug-drug' interaction occurs because the first drug (the inducer) greatly changes the rate at which the second drug (CYP3A4 substrate) is removed from the body. Many drugs increase CYP3A4 activity by binding to a receptor called the Pregnane-X-Receptor (PXR), which is a major switch that controls the expression of the CYP3A4 gene. Using human liver cells we have demonstrated that sulforaphane (SFN), found in broccoli, can block drugs from activating the PXR receptor, thereby inhibiting the switch that causes CYP3A4 induction. The purpose of this project is to determine if SFN can be used to block adverse DDIs that occur when drugs bind to and activate the PXR receptor and subsequently induce CYP3A4 activity. We will recruit 24 human volunteers to participate in the study. This project will determine whether SFN can prevent the drug Rifampin from binding to PXR and increasing CYP3A4 activity in humans following oral administration of SFN (broccoli sprout extract). The rate of removal of a small dose of the drug midazolam will be used to determine the enzymatic activity of CYP3A4 before and following treatment with Rifampin, in the presence or absence of SFN, since midazolam is only eliminated from the bloodstream by CYP3A4. . We predict that SFN will prevent the increase in midazolam clearance (metabolism) that normally follows treatment with the antibiotic, rifampicin.

This research is important because it could potentially lead to a simple, cost-effective way of preventing one of the most common causes of adverse drug-drug interactions that occurs today. For example, rifampicin, which is a cheap and effective antibiotic used to treat TB, cannot be used in HIV/AIDS patients because it increases the metabolism of many of the antiretroviral drugs used to treat HIV/AIDS. TB is a major opportunistic infection in AIDS patients, so this is a serious clinical problem, especially in developing countries where more expensive alternative drug therapies are not available. We hypothesize that co-formulation of rifampicin with SFN could block this drug-drug interaction without altering its efficacy, thereby allowing its use in HIV/AIDS patients infected with TB. This is but one example of numerous drug-drug interactions that occur via this mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Adults from all ethnicities will be encouraged to participate, with our recruitment efforts we expect similar profile as that of the greater Seattle area.

Exclusion Criteria:

Exclusion criteria address a mix of medical and practical issues and include:

* Medical history of gastrointestinal, hepatic, or renal disorders
* Pregnancy or lactation
* Known allergies/intolerances to any foods used in the feeding trial
* Weight loss or gain greater than 4.5 kg within the past year
* Major changes in eating habits within the past year (e.g. adoption of a faddish diet)
* Antibiotic use within the past 3 months
* Body weight greater than 150% of desirable
* Exercise patterns that require or result in major changes in diet
* Current use of prescription medication (including oral contraceptives)
* Current use of over-the-counter medications and herbal supplements
* Regular exposure to passive smoke
* Occupational exposure to smoke or organic solvents
* Food dislikes that would preclude participation in the feeding trial
* Alcohol intake of greater than 2 drinks/day (2 drinks=720 mL beer, 240 mL wine, or 9 mL spirits). Additionally, before the trial, participants will have a blood draw to be sent to the UW Medical Center Lab for liver and kidney functions profile and pregnancy test for women. Those with abnormal test results will be excluded as well as pregnant women.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2008-03; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L Eaton, PhD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - UW General Clinical Research Center, Seattle, Washington

REFERENCES:
- [Background] Poulton EJ, Levy L, Lampe JW, Shen DD, Tracy J, Shuhart MC, Thummel KE, Eaton DL. Sulforaphane is not an effective antagonist of the human pregnane X-receptor in vivo. Toxicol Appl Pharmacol. 2013 Jan 1;266(1):122-31. doi: 10.1016/j.taap.2012.10.029. Epub 2012 Nov 12. PMID 23153560

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 29 participants signed consent form. 23 participants had full measures for data analysis.
Groups:
- Cross-over Trial -Sequence ABC: Three-armed, randomized, crossover trial, 7 days each arm. Arm A: 450 μmol SFN (Broccoli Sprout extract) and Rifampin, then Arm B: 450 μmol SFN (Broccoli Sprout extract), then Arm C: Placebo and Rifampin
- Sequence ACB: Three-armed, randomized, crossover trial, 7 days each arm. Arm A: 450 μmol SFN (Broccoli Sprout extract) and Rifampin then Arm C: Placebo and Rifampin and then Arm B: 450 μmol SFN (Broccoli Sprout extract)
- Sequence BAC: Three-armed, randomized, crossover trial, 7 days each arm. Arm B: 450 μmol SFN (Broccoli Sprout extract) then Arm A: 450 μmol SFN (Broccoli Sprout extract) and Rifampin and then Arm C: Placebo and Rifampin
- Sequence BCA: Three-armed, randomized, crossover trial, 7 days each arm. Arm B: 450 μmol SFN (Broccoli Sprout extract), then Arm C: Placebo and Rifampin, and then Arm A: 450 μmol SFN (Broccoli Sprout extract) and Rifampin
- Sequence CAB: Three-armed, randomized, crossover trial, 7 days each arm. Arm C: Placebo and Rifampin, then Arm A: 450 μmol SFN (Broccoli Sprout extract) and Rifampin and then Arm B: 450 μmol SFN (Broccoli Sprout extract)
- Sequence CBA: Three-armed, randomized, crossover trial, 7 days each arm. Arm C: Placebo and Rifampin, then Arm B: 450 μmol SFN (Broccoli Sprout extract), and then Arm A: 450 μmol SFN (Broccoli Sprout extract) and Rifampin
Period: Overall Study
Arm/Group | Cross-over Trial -Sequence ABC | Sequence ACB | Sequence BAC | Sequence BCA | Sequence CAB | Sequence CBA
Started | 6 | 4 | 5 | 6 | 4 | 4
Completed | 4 | 4 | 4 | 5 | 3 | 3
Not Completed | 2 | 0 | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cross-Over Trial: Crossover trial, three-armed, randomized. The PXR ligand rifampicin (300 mg/d)was given alone for 7 days in Arm 1, or in daily combination with 450 μmol SFN (Broccoli Sprout extract) in Arm 2; SFN was given alone in arm 3. 29 participants consented, analysis done on 23 who finished all arms.
Arm/Group | Cross-Over Trial
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.7 (3.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 23
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Midazolam Clearance (Pharmacokinetic Measure of Cytochrome P450 3A4 Activity)
Time Frame: 7 days
Measure: Mean (Standard Deviation); unit: ng*min/ml
Groups:
- Rifampicin Alone: Subjects are given 300 mg / 7 days of rifampicin to induce CYP3A4. Midazolam clearance is measured on the 8th day. Rifampicin: Rifampicin, an antibiotic used to treat TB, is administered at a dose of 300 mg day x 7 days to induce CYP3A5.
- Broccoli Sprout Extract Plus Rifampin: Sulforaphane (SFN), a natural product derived from broccoli sprouts, is utilized as a putative inhibitor of ligand (Rifampin) activation of the Pregnane X-receptor. In this arm, both SFN (putative inhibitor of ligand binding to PXR) and Rifampin (strong activating ligand of PXR) are given together.
  sulforaphane plus rifampicin: Sulforaphane (SFN) is an isothiocyanate derived from the plant phytochemical, glucoraphinin. It appears to inhibit ligand binding to the ligand activated nuclear transcription factor, Pregnane X-Receptor (PXR). This arm tests the hypothesis that SFN can block ligand binding to the PXR, thereby inhibiting transcriptional activation of PXR-regulated genes. Sulforaphane is administered daily for 7 days as a broccoli sprout extract, at a dose rate of 75 mg (~420 umoles)per day for 7 days. Rifampicin is also administered once per day at a dose rate of 300 mg/day for 7 days.
- Broccoli Sprout Extract Alone: This arm involves the administration of Sulforaphane (SFN) alone, in the absence of the PXR ligand, rifampicin. The hypothesis is that SFN will have no effect on the expression of PXR-regulated genes. Alternatively, it is possible that SFN could inhibit as yet unidentified endogenous ligands to the PXR receptor, thereby causing down-regulations of genes regulated wholely or in part by PXR. SFN is administered as a broccoli sprout extract at a dose rate of 75 mg (~420 umoles) per day for 7 days.
  sulforaphane alone: Sulforaphane (SFN) is an isothiocyanate derived from the plant phytochemical, glucoraraphinin. It appears to inhibit ligand binding to the ligand activated nuclear transcription factor, Pregnane X-Receptor (PXR). This arm tests the hypothesis that SFN can block ligand binding to the PXR, thereby inhibiting transcriptional activation of PXR-regulated genes
Arm/Group | Rifampicin Alone | Broccoli Sprout Extract Plus Rifampin | Broccoli Sprout Extract Alone
Number analyzed (Participants) | 23 | 23 | 23
ng*min/ml
  MDZ AUC Day 1 | 604 (212) | 552 (171) | 541 (222)
  MDZ AUC Day 8 | 156 (72) | 135 (70) | 558 (134)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 7 weeks.
Groups:
- Cross-over Trial: Randomized, crossover trial. 1: Rifampicin (300 mg/d) given alone for 7 days; 2: daily combination with 450 μmol SFN (Broccoli Sprout extract); 3: SFN alone. 29 participants consented. The powdered broccoli extract imparted a bitter taste to the cheese soup used as vehicle. We had all potential participants try the soup before committing to participate. 3 participants who initially did not object to the taste did dropout and did not finish any of the study arms due to dislike or intolerance of the extract. Two of these participants became nauseated, one also had vomiting but it was determined that the subject was suffering from the flu and thus the response was deemed by our attending physician not to be solely treatment related. Three additional participants did not complete all their study periods (one developed apparent lactose intolerance to the soup, one did not routinely comply with study activities, and one relocated out of state after the second study period).
Arm/Group | Cross-over Trial
Serious Adverse Events (participants affected / at risk) | 0/29
Other Adverse Events (participants affected / at risk) | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No